CLINICAL TRIAL: NCT05068739
Title: Needle Knife Fistulotomy Versus Partial Ampullary Endoscopic Mucosal Resection for Difficult Biliary Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Collaborators: Cukurova University (Other)
Responsible Party: Principal Investigator, Salih Tokmak, Asisstant Professor, Duzce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKF vs. PA-EMR
Record Dates: First submitted 2021-09-20; First posted 2021-10-06 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Biliary Disease; Common Bile Duct Calculi; Biliary Stricture; Malignant Hepatobiliary Neoplasm; Pancreatic Disease
Keywords: ERCP; cannulation; endoscopic sphincterotomy
MeSH Terms: conditions — Gallbladder Diseases; Gallstones; Pancreatic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PA-EMR (Partial ampullary endoscopic mucosal resection) (Experimental): Partial ampullary endoscopic mucosal resection
  Interventions: Procedure: PA-EMR
- NKF(Needle knife fistulotomy) (Active Comparator): Needle knife fistulotomy
  Interventions: Procedure: NKF

INTERVENTIONS:
Procedure: PA-EMR — Standard oval-shaped, braided wire polypectomy snare with 10 mm or 20 mm loop diameter will be used. With the duodenoscope in a semi-long position, the tip of the snare will be anchored just below the transverse fold of the ampulla and opened above-downwards fashion until the orifice will be seen. The orifice will be strictly preserved to avoid the risk of PEP and approximately the upper two-thirds of the ampullary mound will be grabbed by the snare. The direction and the depth will be controlled by combined movements of the elevator and wheels of the duodenoscope. After removal of the mucosa, the wall of choledochus will be seen clearly and standard wire-guided cannulation (WGC) will be performed. If cannulation can not be achieved with WGC, an additional incision will be performed to the wall of the choledochus with a needle knife.
  Arms: PA-EMR (Partial ampullary endoscopic mucosal resection)
Procedure: NKF — The needle knife will be placed at the junction of the upper one-third and lower two-thirds of the papillary roof (bulging portion). Minimal, superficial incisions will be made in the 11-12 o'clock direction. The length of the fistulotomy will be at the endoscopist's discretion, depending on the shape of the papilla. The cut will be extended until bile juice, the pinkish bile duct mucosa, and/or the bulging of the white sphincter of the Oddi's muscle is visible.
  Arms: NKF(Needle knife fistulotomy)

SUMMARY:
The aims of this study are to compare the needle knife fistulotomy (NKF) technique versus the partial ampullary endoscopic mucosal resection (PA-EMR) technique in patients with difficult biliary cannulation and to assess the incidence rate of complications between these cannulation methods.

DETAILED DESCRIPTION:
Cannulation success with standard techniques reported to be around 95% even in expert hands and despite all efforts, it can be challenging that needs an alternate intervention.

NKF is recommended as the initial technique for pre-cutting because the rate of post-ERCP pancreatitis (PEP) is significantly low but there is an ongoing debate about limiting its use in certain types of papillae with a long intra-mural segment

Indeed the shape of the papillae influences the success of bile duct cannulation and the choice of the pre-cutting technique. Type-2 and Type-3 papillae are more difficult to cannulate than Type-1. NKF can be performed as the initial technique for pre-cutting in protruded Type-2 and Type-3 papillae but it has some limitations.

First of all, the incision can be erratic because it is performed without a guidewire and uncontrolled. This can cause a tattered mucosa as the incision progress and the papillae lose anatomic contours. Some amount of bleeding may also unavoidably occur and the field of view further impaired. If the initial incision line is incorrect and additional incision is needed, more crumpled and deformed papillae with irregular margins may be encountered. These undesired results are frequently experienced and prevent a clean-cut, thus further complicate the cannulation. Even perforation can occur.

Recently the investigators described a novel technique, PA-EMR, for difficult biliary cannulation in patients with protruded Type-2, Type-3, and shar-pei papilla. The investigators hypothesized that with this new technique cannulation success will be higher, procedure time will be shorter and the adverse events will be lower versus NKF technique.

ELIGIBILITY:
Inclusion Criteria:

* Patient who submitted a written informed consent for this trial, and aged between 18-90 years old
* Patient who have naïve papilla (no previous procedure was performed at ampulla)
* Patient who is suspected to have a biliary obstruction or biliary disease
* Patient who is needed to have endoscopic retrograde cholangiopancreatography for treatment of biliary obstruction
* Patient who have risks of post-endoscopic retrograde cholangiopancreatography p

Exclusion Criteria:

* Patient who is pregnant
* Patient with mental retardation
* Patient allergic to contrast agents
* Patient who received sphincterotomy or pancreatobiliary operation previously
* Patient who have ampulla of Vater cancer
* Patient who have difficulty for the approach to ampulla due to abdominal surgery including stomach cancer with Billroth II anastomosis
* Patient who have pancreatic diseases as bellow (at least one more);

  * acute pancreatitis within 30days before enrollment
  * idiopathic acute recurrent pancreatitis
  * pancreas divisum
  * obstructive chronic pancreatitis
  * pancreatic cancer
* Patients with Type-1, non-protruding Type-2 and Type-4 papilla

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Success rate of cannulation | 1 day
  Successful bilary cannulation, verified by fluoroscopic images of correct guidewire positioning in the CBD, and contrast media.

SECONDARY OUTCOMES:
Incidence rate of complications | 1 week
  The rate of complications (if any occur)
Cannulation time | 1 day
  Time from first contact with cannula to papillae to deep cannulation
Procedure time | 1 day
  Total procedure time

CONTACTS AND LOCATIONS:
Overall Officials: Salih Tokmak, Assist. prof, Study Director — Duzce University
Locations (1):
- Duzce University School of Medicine, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Testoni PA, Mariani A, Aabakken L, Arvanitakis M, Bories E, Costamagna G, Deviere J, Dinis-Ribeiro M, Dumonceau JM, Giovannini M, Gyokeres T, Hafner M, Halttunen J, Hassan C, Lopes L, Papanikolaou IS, Tham TC, Tringali A, van Hooft J, Williams EJ. Papillary cannulation and sphincterotomy techniques at ERCP: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2016 Jul;48(7):657-83. doi: 10.1055/s-0042-108641. Epub 2016 Jun 14. PMID 27299638
- [Background] Haraldsson E, Lundell L, Swahn F, Enochsson L, Lohr JM, Arnelo U; Scandinavian Association for Digestive Endoscopy (SADE) Study Group of Endoscopic Retrograde Cholangio-Pancreaticography. Endoscopic classification of the papilla of Vater. Results of an inter- and intraobserver agreement study. United European Gastroenterol J. 2017 Jun;5(4):504-510. doi: 10.1177/2050640616674837. Epub 2016 Oct 17. PMID 28588881
- [Background] Katsinelos P, Lazaraki G, Chatzimavroudis G, Zavos C, Kountouras J. The endoscopic morphology of major papillae influences the selected precut technique for biliary access. Gastrointest Endosc. 2015 Apr;81(4):1056. doi: 10.1016/j.gie.2014.11.018. No abstract available. PMID 25805488
- [Background] Sriram PV, Rao GV, Nageshwar Reddy D. The precut--when, where and how? A review. Endoscopy. 2003 Aug;35(8):S24-30. doi: 10.1055/s-2003-41528. No abstract available. PMID 12929050